CLINICAL TRIAL: NCT04458116
Title: Curcumin Supplementation Effects on Markers of Cardiovascular Risk, Inflammation, Oxidative Stress and Functional Capacity in Patients With Coronary Arterial Disease
Brief Title: Effects of Curcumin on Markers of Cardiovascular Risk in Patients With CAD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We could not start the project
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Denise Mafra9
Record Dates: First submitted 2020-05-28; First posted 2020-07-07 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease; Oxidative Stress; Inflammation
Keywords: Coronary Artery Disease; Curcumin; Oxidative Stress; Inflammation
MeSH Terms: conditions — Coronary Artery Disease; Inflammation | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: Is a longitudinal randomized clinical study where participants will be randomized into two groups: Turmeric Group, in which participants will receive 1.5 grams of turmeric 95% curcumin (ACTIVE PHARMACEUTICA LTDA) for 1 month (3 capsules / day containing 500mg each for 4 weeks), and placebo group, where participants will receive capsules containing corn starch. Randomization will be done in blocks.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tumeric Group (Experimental): participants will receive capsules containing 1.5 grams of turmeric 95% curcumin
  Interventions: Dietary Supplement: Curcumin
- Placebo Group. (Placebo Comparator): will receive capsules containing corn starch.
  Interventions: Dietary Supplement: Curcumin

INTERVENTIONS:
Dietary Supplement: Curcumin — Participants will receive 1.5 grams of turmeric 95% curcumin for 1 month (3 capsules / day containing 500mg each for 4 weeks).

SUMMARY:
- General Objective To evaluate the effects of curcumin supplementation on cardiovascular risk markers, inflammation, oxidative stress and functional capacity in participants with coronary artery disease.

Specific Objectives

Assess, before and after supplementation with turmeric:

* The nutritional status of the participants;
* Blood pressure;
* Atherogenic risk;
* The expression of transcription factors (Nrf2 and NF-kB), antioxidant enzymes (NQO1, HO-1, sirtuin 1 (SIRT-1)), NLPR3 receptor, as well as the levels of inflammatory cytokines (IL-6, tumor necrosis factor-alpha (TNF-α), protein C reactive (PCR), IL-1, IL 18) and vascular cell adhesion protein 1 (VCAM-1) and E-selectin adhesion molecules;
* Routine biochemical parameters;
* Lipid peroxidation and oxidized LDL;
* The 6-minute walk test, the recovery heart rate and the chair lift test;
* Modifiable risk factors before and after supplementation;
* The comparison of all parameters between groups.

DETAILED DESCRIPTION:
Coronary Artery Disease (CAD) is the leading cause of death worldwide. CAD refers to the pathological process of atherosclerosis that affects the coronary arteries, often leading to obstruction by an atheromatous plaque. Oxidative stress is one of the most potent inducers of vascular inflammation in atherogenesis. Reactive oxygen species (ROS) regulate through nuclear factor kB (NF-kB), transcription factors and genes related to inflammation, thus, activation of NF-kB by ROS in the atherosclerosis patient is associated with vascular dysfunction and thus with inflammation and atherosclerosis. Recently, researchers have discovered a transcription factor identified as nuclear factor-erythroid 2-related factor 2 (Nrf2) transcription factor, which is responsible for the expression of antioxidant response element genes that can inhibit this pathway, thus providing cellular protection. Thus, several nutritional strategies have been studied, including the use of curcumin, a chemical compound of the class of curcumin produced by turmeric root (Curcuma longa). Turmeric is capable of promoting the activation of nuclear factor-erythroid 2-related factor 2 (Nrf2) transcription factor and inflammasome (NLPR3). These factors, in turn, are involved with the activity of nuclear factor kappa-B (NF-kB), a transcription factor that increases the synthesis of inflammatory cytokines. Thus, the present study aims to evaluate the effects of turmeric supplementation on cardiovascular risk markers, inflammation, oxidative stress and evaluation of functional capacity. Perspectives: This study aims to improve the inflammatory and oxidative stress status of patients with CAD with the use of turmeric, and thus try to reduce the risk factors related to the onset and progression of coronary artery disease.

ELIGIBILITY:
Inclusion criteria:

* Non-smokers
* with a previous diagnosis of coronary artery disease and / or altered myocardial scintigraphy, both performed by a cardiologist.

Exclusion criteria:

* autoimmune and infectious diseases
* pregnant and lactating women
* cancer
* AIDS;
* participants using catabolic drugs, antioxidant vitamin supplements and habitual intake of turmeric and turmeric.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-10 (Estimated); Primary Completion 2021-05-10 (Estimated); Study Completion 2021-05-10 (Estimated)

PRIMARY OUTCOMES:
The effects of curcumin supplementation on the expression of transcription factors | 4 months
  Get blood samples to evaluate the supplementation effects in antioxidants biomarkers- nuclear receptor factor 2 (Nrf2), glutathioneperoxidase (GPx), heme oxygenase-1 (HO-1)
The effects of curcumin supplementation on antioxidant enzymes. | 4 months
  Get blood samples to evaluate the supplementation effects in antioxidants biomarkers glutathioneperoxidase (GPx), heme oxygenase-1 (HO-1), NQO1
The effects of curcumin supplementation on inflammatory cytokines. | 4 months
  Get blood samples to evaluate the supplementation effects on cytokines

SECONDARY OUTCOMES:
The effects of curcumin supplementation on blood pressure | 4 months
  Measurement of blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Denise Mafra, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No